CLINICAL TRIAL: NCT05181813
Title: Clinical Evaluation of Calcium Hydroxide Mixed With Gingerols Versus Metapex in Treatment of Primary Teeth With Infected Necrotic Pulp
Brief Title: Treatment of Infected Pulp in Primary Teeth With a Mixture of Calcium Hydroxide and Gingerols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Fathi Abdulraqeb Qasem, PhD in Pediatric Dentistry, Pediatric Dentistry Department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06030718
Record Dates: First submitted 2021-11-30; First posted 2022-01-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Primary Teeth; Pulp Necroses; Infected Pulp; Root Canal Treatment
Keywords: Pediatric Dentistry; Pulpectomy; Infected Pulp; Necrotic Pulp; Gingerols; Calcium Hydroxide; Metapex; Ginge-Cal
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Metapex

STUDY DESIGN:
Intervention Model Description: Selected children will be divided randomly into 2 groups:
  Group 1: Ginge-Cal group: primary molars were filled with a creamy mixture of pulpectomy paste of Gingerols and Calcium Hydroxide.
  Group 2: Metapex group: primary molars were filled with a ready-made injectable creamy mixture pulpectomy paste of Metapex.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Ginge-Cal group: (Experimental): primary molars were filled by creamy mixture pulpectomy paste of Gingerols and Calcium Hydroxide.
  Interventions: Procedure: Ginge-Cal
- Group 2: Metapex group (Active Comparator): primary molars were filled by a ready-made injectable creamy mixture pulpectomy paste of Metapex
  Interventions: Procedure: Metapex

INTERVENTIONS:
Procedure: Ginge-Cal — Fill the infected root canal of of primary teeth with Gingerols extract and Calcium Hydroxide (Ginge-Cal)
  Arms: Group 1: Ginge-Cal group:
Procedure: Metapex — Fill the infected root canal of of primary teeth with Metapex
  Arms: Group 2: Metapex group

SUMMARY:
This study was conducted to evaluate Calcium Hydroxide mixed with Gingerols versus Metapex in treatment of primary teeth with infected necrotic pulp

DETAILED DESCRIPTION:
Study compare Calcium Hydroxide mixed with Gingerols versus Metapex in treatment of primary teeth with infected necrotic pulp clinically and radiographically

ELIGIBILITY:
Inclusion Criteria:

1. The cooperation of the child and parents, during the treatment plan, and the commitment to attend the follow-up appointments.
2. Parents signed the consent to participate in the study.
3. Absence of any systemic disease, which would contraindicate pulp therapy.
4. Child didn't have any history of a sensitive reaction to any component of used materials.
5. Present half to two third of tooth root or more
6. Root with signs or symptoms of infected necrotic pulp or chronic abscess, with or without sinus tract, soft tissue swelling, mobility or tenderness to percussion, and internal or external root resorption or unsuccessful past pulp treatment.

Exclusion Criteria:

All that does not correspond to inclusion criteria.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage of primary teeth with control necrotic pulp by clinical examination | Up to 18 months
  The primary outcome was evaluated using clinical evaluation methods. Two pediatric dentists who are blind to treated teeth will conduct the clinical evaluation. A third examiner will be consulted if there is a disagreement between the results of the first two. Clinical success will be judged to have occurred when there are no reports of pain, abscess, fistula, or mobility inconsistent with chronological age.
Percentage of primary teeth with control necrotic pulp by radiographic examination | Up to 18 months
  The primary outcome was evaluated using Radiographic evaluation methods. Two pediatric dentists who are blind to treated teeth will conduct the clinical evaluation. A third examiner will be consulted if there is a disagreement between the results of the first two. Radiographic success will be evidenced by a decrease or absence of periapical or furcation area radiolucency and pathological root resorption

CONTACTS AND LOCATIONS:
Overall Officials: Fathi A Qasem, PhD, Principal Investigator — Assistant Professor of Pediatric Dentistry Faculty of Dentistry Thamar University Yemen; Salwa M Awad, Prof, Study Director — Prof. of Pediatric Dentistry and Dental Public Health Faculty of Dentistry Mansoura University; Rizk A ELagamy, PhD, Study Director — Lecturer of Pediatric Dentistry Faculty of Dentistry Mansoura University
Locations (1):
- Faculty of Dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol to other researchers
Supporting Information: Study Protocol
Time Frame: Within 6 Months
Access Criteria: For anyone

REFERENCES:
- [Derived] Qasem FA, Awad SM, Elagamy RA. Effectiveness of Calcium Hydroxide and Gingerols Mixture as a Novel Obturation Material for Infected Root in Primary Teeth: A Randomized Clinical Trial. Int J Dent. 2024 Feb 8;2024:5528260. doi: 10.1155/2024/5528260. eCollection 2024. PMID 38362239